CLINICAL TRIAL: NCT02767570
Title: Personalized Gait Training With Feedback to Reduce Knee Pain From Osteoarthritis
Brief Title: Long-Term Effectiveness of Walking Training in Patients With Knee Osteoarthritis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study data collection was terminated due to COVID-19 pandemic and will not resume.
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: O1811-R
Record Dates: First submitted 2016-05-04; First posted 2016-05-10 (Estimated); Results first posted 2022-04-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-02

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis, Knee; Arthritis; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee; Arthritis; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gait Training; Altered Foot Progression Angle (Experimental): Participants will receive personalized gait training while walking on a treadmill with real-time, haptic feedback. The goal of the training is to encourage participants to adopt an altered foot progression angle in an attempt to alter the distribution of forces crossing the knee joint. Training will occur once a week for six weeks. This will be followed by a 46-week home and community-based walking program to practice and internalize the new personalized, gait pattern and to encourage daily walking. Refresher training with haptic feedback will be offered at weeks 11, 25 and 39 to enhance internalization of the new foot progression angle.
  Interventions: Other: Gait Training; Altered Foot Progression Angle
- Gait Training; Consistent Foot Progression Angle (Experimental): Participants will receive personalized gait training while walking on a treadmill with haptic feedback. The goal of the training is to encourage participants to maintain a consistent foot progression angle in an attempt to minimize the variability in the forces crossing the knee joint. Training will occur once a week, for 6 weeks. This will be followed by a 46-week home and community-based walking program to encourage daily walking. Refresher training with haptic feedback will be offered at weeks 11, 25 and 39 to maintain foot progression angle consistency.
  Interventions: Other: Gait Training; Consistent Foot Progression Angle

INTERVENTIONS:
Other: Gait Training; Altered Foot Progression Angle — Participants will receive personalized gait training while walking on a treadmill with real-time, haptic feedback to encourage them to adopt a new foot progression angle. Participants will walk for an additional ten minutes per day to internalize their new foot progression angle over 52 weeks.
  Arms: Gait Training; Altered Foot Progression Angle
Other: Gait Training; Consistent Foot Progression Angle — Participants will receive personalized gait training while walking on a treadmill with haptic feedback to encourage them to maintain a consistent foot progression angle. Participants will walk an additional ten minutes per day to internalize the consistency of their foot progression angle over 52 weeks.
  Arms: Gait Training; Consistent Foot Progression Angle

SUMMARY:
Nearly one out of every two Americans will develop knee osteoarthritis by age 85. Over 20 million Americans, including nearly three million Veterans, currently have painful knee arthritis that limits their daily activity or recreation. The vast majority of those individuals will be prescribed anti-inflammatory drugs that provide some pain relief but do not slow the progression of the disease. Often people with knee arthritis are told they must live with the pain until they become appropriate candidates for knee replacement surgery, but that can require tolerating the pain and limiting function for many years. Because of other health issues, some individuals are never acceptable surgery candidates. What is desperately needed are better conservative approaches for treating these patients. Two such approaches will be tested and compared in this study.

DETAILED DESCRIPTION:
This study is a randomized controlled trial to investigate conservative treatments for individuals with painful knee osteoarthritis (OA). The study will recruit participants who have isolated, medial compartment knee OA. Subjects will be assigned to one of two gait training groups. Both groups will undergo gait analysis to determine their foot progression angle at their comfortable walking speed. Both groups will receive personalized gait retraining to either alter their foot progression angle or to achieve consistency of their natural foot progression angle.

Gait retraining will consist of once a week sessions for six weeks. The gait training will use a fading feedback approach, where the percentage of each weekly session during which feedback is used is decreased from week to week until no feedback is used by the last training session. Throughout the six-week training period subjects will be encouraged to practice their gait for at least ten minutes per day. Subjects will continue to practice their gait throughout the remainder of the 52-week intervention. Subjects will have their walking activity recorded using a 3-axis pedometer. Compared to their baseline walking activity, participants will be instructed to increase their daily walking by ten minutes per day throughout the 52-week intervention.

All subjects will receive monthly phone calls to encourage maintaining a regular walking regimen. Walking activity will be monitored periodically using a pedometer. Subjects will receive knee MRIs and weight-bearing knee radiographs at the start and end of the study. All participants will complete pain evaluations and clinical knee score questionnaires during the study. The investigators expect that subjects in both groups will have a reduction in knee pain over the course of the 52-week intervention. The primary objective of the study it to determine if the change in pain between baseline and week 52 is different between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with isolated, medial compartment knee OA of at least six months duration
* Kellgren-Lawrence grade of I, II, or III
* Age greater than 18 years at the time of enrollment
* Ability to give informed consent
* Knee pain more than three days per week on average
* Average knee pain in medial compartment between 3 and 9 on an 11-point Numerical Rating Scale, and greater than pain in other compartments
* Ambulatory without aids
* Able to walk for at least 25 consecutive minutes
* Able to walk on treadmill safely at 0.7 m/s or faster
* Able to reduce the prominent peak of the knee adduction moment by changing foot progression angle

Exclusion Criteria:

* Body mass index equal to or greater than 35
* Pregnancy
* Plans for knee replacement within the next 12 months
* Contraindications to MRI
* Nerve or muscle disease associated with walking difficulty
* Narcotic pain medication usage
* History of rheumatoid arthritis or autoimmune disease
* An episode of gout or pseudogout in the knee in the past year
* History of neuropathic arthropathy, infectious disease, or other major systemic diseases
* Current or recent past use (within two months) of oral corticosteroids
* Cognitive impairments that would limit a subject's understanding
* Expecting a significant change in activity level or weight within the next 12 months
* Regularly participates in high impact activities such as running, soccer, basketball, etc.
* Unable to perform the 3rd stage of the 4-stage balance test, which involves holding a tandem stance for 10 seconds

The following criteria apply only to the affected osteoarthritic limb:

* History of symptomatic arthritis in lower limb joints other than the knees that is more severe than knee arthritis
* Replacement of any lower extremity joint
* Lateral tibiofemoral joint space width less than medial
* Recurrent giving way of the knee
* Symptoms arising primarily from a meniscal or ligament pathology or other structure not directly related to osteoarthritis as identified by physical exam, health record, or MRI
* Symptoms originating primarily from the patellofemoral joint
* Avascular necrosis
* Recent (within two months) knee injury or surgery
* Planned use of hinged knee brace in next 12 months
* Severe knee malalignment of more than 10 degrees from neutral
* Intra-articular injection within the past 2 months or planned for the next 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Kolesar, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (2):
- United States (2):
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - Stanford University, Depts: Bioengineering; Orthopaedics, Stanford, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Uhlrich SD, Mazzoli V, Silder A, Finlay AK, Kogan F, Gold GE, Delp SL, Beaupre GS, Kolesar JA. Personalised gait retraining for medial compartment knee osteoarthritis: a randomised controlled trial. Lancet Rheumatol. 2025 Oct;7(10):e708-e718. doi: 10.1016/S2665-9913(25)00151-1. Epub 2025 Aug 12. PMID 40816302

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via clinician referrals, approved searches of medical record databases, and advertisements in print media and online. The first participant was enrolled in August 2016 and the last participant was enrolled in June 2019.
Pre-assignment Details: Interested individuals were initially screened via telephone or web-based questionnaire. Eligible individuals then underwent an in-person screen to confirm the location and severity of knee pain. Anterior-posterior weightbearing radiographs were obtained and given a KL grade. Participants who met the radiographic inclusion criteria were invited to the motion laboratory for a gait assessment. Those who were able to reduce their KAM peak by at least 5% with an FPA modification were randomized.
Period: Overall Study
Arm/Group | Gait Training; Altered Foot Progression Angle | Gait Training; Consistent Foot Progression Angle
Started | 34 | 34
Per Protocol Week 6 | 31 | 33
Completed | 25 | 24
Not Completed | 9 | 10
Not completed — Lost to Follow-up | 3 | 0
Not completed — COVID shutdown | 2 | 5
Not completed — Increased pain | 2 | 0
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Unrelated medical issue | 1 | 1
Not completed — Received intra-articular injection | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gait Training; Altered Foot Progression Angle | Gait Training; Consistent Foot Progression Angle | Total
Number analyzed (Participants) | 34 | 34 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.32 (7.66) | 64.53 (7.63) | 64.43 (7.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 41
  Male | 13 | 14 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 34 | 34 | 68
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 6 | 10
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 0 | 1 | 1
  White | 28 | 26 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34 | 34 | 68
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.53 (3.26) | 27.37 (3.95) | 26.45 (3.71)
Kellgren-Lawrence classification of knee OA [Count of Participants; unit: Participants] — Classification of knee OA using 5 grades ranging from 0 (no presence of OA) to 4 (severe OA)
  Participants
    Grade 1 | 7 | 7 | 14
    Grade 2 | 14 | 17 | 31
    Grade 3 | 13 | 10 | 23
NRS pain, medial [Mean (Standard Deviation); unit: units on a scale] — Medial compartment knee pain assessed using an 11-point numeric rating scale (NRS) ranging from 0 (no pain) to 10 (worst pain imaginable).
  units on a scale | 4.32 (1.32) | 4.00 (1.21) | 4.16 (1.27)
KAM peak, natural FPA [Mean (Standard Deviation); unit: %Bodyweight*Height] — Peak knee adduction moment (KAM), a surrogate measure for medio-lateral load distribution in the knee, measured when walking with a natural foot progression angle (FPA). A reduction in KAM indicates a shift in loading from the medial to the lateral compartment of the knee.
  %Bodyweight*Height | 3.25 (1.05) | 3.30 (1.05) | 3.27 (1.04)
KAM peak, target FPA [Mean (Standard Deviation); unit: %Bodyweight*Height] — Peak knee adduction moment (KAM), a surrogate measure for medio-lateral load distribution in the knee, measured when walking with the target foot progression angle (FPA). A reduction in KAM indicates a shift in loading from the medial to the lateral compartment of the knee.
  %Bodyweight*Height | 2.87 (1.05) | 3.30 (1.05) | 3.08 (1.06)
WOMAC pain [Mean (Standard Deviation); unit: units on a scale] — Pain subscale score of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), a self-report questionnaire to evaluate knee OA. The possible score range for the Pain subscale is 0-20. The raw scores were then normalized to a range of 0-100, with higher scores indicating worse pain.
  units on a scale | 70.74 (12.86) | 71.21 (11.18) | 70.97 (11.97)
WOMAC function [Mean (Standard Deviation); unit: units on a scale] — Physical Function subscale score of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), a self-report questionnaire to evaluate knee OA. The possible score range for the Physical Function subscale is 0-68. The raw scores were then normalized to a range of 0-100, with higher scores indicating worse function.
  units on a scale | 75.74 (14.23) | 73.17 (13.06) | 74.45 (13.62)
Daily steps [Mean (Standard Deviation); unit: steps/day] — Daily steps measured and averaged over one week using a pedometer carried by the participant.
  steps/day | 6343 (2678) | 6280 (3073) | 6311 (2860)

OUTCOME MEASURES:

1. Primary Outcome: Change in Medial Knee Pain
Description: Change in medial knee pain between baseline and week 52 using an 11-point Numeric Rating Scale (NRS) to assess average medial knee pain over the past 7 day period. Possible scores range from 0 (no pain) to 10 (worst pain imaginable). Change = (Week 52 score - Baseline score).
Time Frame: Baseline and Week 52
Population: Intent-to-treat population. Missing data were imputed using the Markov chain Monte Carlo method for continuous variables.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gait Training; Altered Foot Progression Angle | Gait Training; Consistent Foot Progression Angle
Number analyzed (Participants) | 34 | 34
score on a scale | -2.5 (2.2) | -1.3 (2.3)
Statistical Analysis 1: Comparison: Gait Training; Altered Foot Progression Angle vs Gait Training; Consistent Foot Progression Angle; For the primary hypothesis that there would be a greater reduction in pain for the altered compared to the consistent FPA group, an effect size of 0.57 was assumed. To achieve 80% power with an alpha of 0.05, 39 participants per group were needed, so our recruitment goal was 40 subjects per group; Test type: Superiority; p = 0.001, Regression, Linear — The threshold for statistical significance was p=0.05; Mean Difference (Net) = -1.2, 95% CI 2-sided [-1.9 to -0.5] — Difference = Altered FPA - Consistent FPA

2. Primary Outcome: Change in Knee Adduction Moment
Description: Change in magnitude of the more prominent peak in the knee adduction moment (KAM), a surrogate measure for medio-lateral load distribution in the knee, between baseline and week 52. A reduction in KAM indicates a shift in loading from the medial to the lateral compartment of the knee. Change = (Week 52 - Baseline).
Time Frame: Baseline and Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: %Bodyweight*Height
Arm/Group | Gait Training; Altered Foot Progression Angle | Gait Training; Consistent Foot Progression Angle
Number analyzed (Participants) | 34 | 34
%Bodyweight*Height | -0.17 (0.47) | 0.08 (0.33)
Statistical Analysis 1: Comparison: Gait Training; Altered Foot Progression Angle vs Gait Training; Consistent Foot Progression Angle; Test type: Superiority; p < 0.001, Regression, Linear — The threshold for statistical significance was p=0.05; Mean Difference (Net) = -0.26, 95% CI 2-sided [-0.39 to -0.13] — Difference = Altered FPA - Consistent FPA

3. Secondary Outcome: Change in Medial T1rho Relaxation Time
Description: Change in T1rho relaxation time measured from quantitative MRI in the medial compartment of the knee between baseline and week 52. T1ρ relaxation time is sensitive to changes in proteoglycan content in the articular cartilage. Increased values of T1rho indicate increased depletion of proteoglycans and increased cartilage degeneration. Change = (Week 52 - Baseline).
Time Frame: Baseline and Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Gait Training; Altered Foot Progression Angle | Gait Training; Consistent Foot Progression Angle
Number analyzed (Participants) | 34 | 34
ms | -1.72 (5.68) | 2.02 (5.53)
Statistical Analysis 1: Comparison: Gait Training; Altered Foot Progression Angle vs Gait Training; Consistent Foot Progression Angle; Test type: Superiority; p = 0.006, Regression, Linear — The threshold for statistical significance was p=0.05; Mean Difference (Net) = -3.74, 95% CI 2-sided [-6.42 to -1.05] — Difference = Altered FPA - Consistent FPA

4. Secondary Outcome: Change in Medial T2 Relaxation Time
Description: Change in T2 relaxation time measured from quantitative MRI in the medial compartment of the knee between baseline and week 52. T2 relaxation time is sensitive to changes in water content and collagen matrix integrity of the articular cartilage. Increased values of T2 indicate increased cartilage degeneration. Change = (Week 52 - Baseline).
Time Frame: Baseline and Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Gait Training; Altered Foot Progression Angle | Gait Training; Consistent Foot Progression Angle
Number analyzed (Participants) | 34 | 34
ms | -0.58 (2.65) | -0.52 (3.11)
Statistical Analysis 1: Comparison: Gait Training; Altered Foot Progression Angle vs Gait Training; Consistent Foot Progression Angle; Test type: Superiority; p = 0.93, Regression, Linear — The threshold for statistical significance was p=0.05; Mean Difference (Net) = -0.06, 95% CI 2-sided [-1.42 to 1.30] — Difference = Altered FPA - Consistent FPA

5. Secondary Outcome: Change in Lateral T1rho Relaxation Time
Description: Change in T1rho relaxation time measured from quantitative MRI in the lateral compartment of the knee between baseline and week 52. T1ρ relaxation time is sensitive to changes in proteoglycan content in the articular cartilage. Increased values of T1rho indicate increased depletion of proteoglycans and increased cartilage degeneration. Change = (Week 52 - Baseline).
Time Frame: Baseline and Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Gait Training; Altered Foot Progression Angle | Gait Training; Consistent Foot Progression Angle
Number analyzed (Participants) | 34 | 34
ms | -1.11 (6.07) | -0.83 (6.80)
Statistical Analysis 1: Comparison: Gait Training; Altered Foot Progression Angle vs Gait Training; Consistent Foot Progression Angle; Test type: Superiority; p = 0.85, Regression, Linear — The threshold for statistical significance was p=0.05; Mean Difference (Net) = -0.29, 95% CI 2-sided [-3.38 to 2.80] — Difference = Altered FPA - Consistent FPA

6. Secondary Outcome: Change in Lateral T2 Relaxation Time
Description: Change in T2 relaxation time measured from quantitative MRI in the lateral compartment of the knee between baseline and week 52. T2 relaxation time is sensitive to changes in water content and collagen matrix integrity of the articular cartilage. Increased values of T2 indicate increased cartilage degeneration. Change = (Week 52 - Baseline).
Time Frame: Baseline and Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Gait Training; Altered Foot Progression Angle | Gait Training; Consistent Foot Progression Angle
Number analyzed (Participants) | 34 | 34
ms | -0.02 (2.14) | -0.02 (1.88)
Statistical Analysis 1: Comparison: Gait Training; Altered Foot Progression Angle vs Gait Training; Consistent Foot Progression Angle; Test type: Superiority; p = 0.99, Regression, Linear — The threshold for statistical significance was p=0.05; Mean Difference (Net) = 0.00, 95% CI 2-sided [-0.89 to 0.90] — Difference = Altered FPA - Consistent FPA

ADVERSE EVENTS:
Description: Death, serious adverse events, and other (non-serious) adverse events were not assessed for the study.
Arm/Group | Gait Training; Altered Foot Progression Angle | Gait Training; Consistent Foot Progression Angle
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Enrollment was lower than expected due to the fact that most interested participants did not meet study inclusion criteria. As a result, we did not reach our pre-specified sample size of 80 participants. In addition, the institutional shutdown due to the COVID-19 pandemic resulted in 7 participants not completing the full 1-year intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/70/NCT02767570/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-29): https://cdn.clinicaltrials.gov/large-docs/70/NCT02767570/ICF_001.pdf